CLINICAL TRIAL: NCT06272617
Title: A Single-center, Single-blind Phase II Clinical Trial of Acupuncture for the Prevention and Treatment of Oral-related Complications Caused by Radiotherapy for Head and Neck Malignant Tumors
Brief Title: Acupuncture for Prevention and Treatment of Oral-related Complications Caused by Radiotherapy for Head and Neck Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: West China Fourth Hospital, Sichuan University (Unknown)
Responsible Party: Principal Investigator, Xingchen Peng, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-960
Record Dates: First submitted 2024-01-30; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Malignant Tumor of Head and/or Neck; Radiotherapy; Complications
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- treatment group (Experimental): verum acupuncture
  Interventions: Device: verum acupuncture
- control group (Sham Comparator): sham acupuncture
  Interventions: Device: sham acupuncture

INTERVENTIONS:
Device: verum acupuncture — a type of acupuncture which is useful
  Arms: treatment group
Device: sham acupuncture — a type of acupuncture which is useless
  Arms: control group

SUMMARY:
A study on the efficacy and safety of acupuncture for the prevention and treatment of oral-related complications caused by radiotherapy for head and neck malignant tumors

DETAILED DESCRIPTION:
The goal of this clinical trial is to investigate the efficacy and safety of acupuncture for oral-related complications in patients with head and neck malignant tumors who receive radiotherapy. The main questions it aims to answer are:

* the efficacy of acupuncture for the prevention and treatment of oral-related complications caused by radiotherapy for head and neck malignant tumors
* the safety of acupuncture for the prevention and treatment of oral-related complications caused by radiotherapy for head and neck malignant tumors

Participants will:

* be treated with real acupuncture or sham acupuncture
* be evaluated to learn the efficacy and safety of acupuncture for the prevention and treatment of oral-related complications caused by radiotherapy for head and neck malignant tumors

Researchers will compare real acupuncture group with sham acupuncture group to see if acupuncture has good efficacy and safety of acupuncture for the prevention and treatment of oral-related complications caused by radiotherapy for head and neck malignant tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with malignant tumors of the head and neck without metastasis
* Age ≥18, ≤80 years old
* ZPS score ≤2
* Receiving radiotherapy alone or concurrent radiotherapy with a radiation dose of >50 Gy, including at least one parotid gland
* Judged to be able to receive acupuncture treatment, with all needle positions identified as accessible
* Signed informed consent form

Exclusion Criteria:

* History of dry mouth, Sjogren's syndrome, or other underlying systemic condition known to cause dry mouth
* Suspected or confirmed physical closure of both salivary gland ducts
* Have a phobia of needles or prohibit the use of acupuncture at any acupuncture points
* Have a history of head and neck radiotherapy
* Have contraindications to acupuncture, including but not limited to bleeding disorders, having skin infections, ulcers or frequent infections
* Have taken any medications or herbs within the past 30 days that may affect salivary function, plan to or eventually take such substances during the study period
* Poor oral hygiene or severe periodontitis
* Poor compliance
* Other patients who, in the opinion of the investigator, are not suitable for participation in this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-07-24 (Estimated); Study Completion 2025-07-24 (Estimated)

PRIMARY OUTCOMES:
Xerostomia questionnaire scores | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Patients self-evaluated xerostomia according to Xerostomia questionnaire(score 0-100);Higher score indicates more severe symptoms

SECONDARY OUTCOMES:
Salivary flow rate | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Researchers-measured unstimulated and stimulated salivary flow rates;Lower value indicates more severe symptoms
Taste function assessed by patients | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Assessed by Patients self-evaluated dysgeusia(score 19-95);Higher score indicates more severe symptoms
Taste function assessed by electrogustometer test | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Assessed by electrogustometer test(score -6 to 34);Higher score indicates more severe symptoms
Taste function assessed by taste strips test | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Assessed by taste strips test(score 0-16);Lower score indicates more severe symptoms
Oral mucositis | 1 week before radiotherapy;twice a week during the treatment(usually every 3 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Oral mucositis is assessed by trained physicians according to World Health Organization (WHO) oral toxicity Scale(grade 1-5);Higher grade indicates more severe symptoms
Dysphagia | 1 week before radiotherapy;at the middle of treatment(3 weeks after the start of radiotherapy);at the end of treatment(the last radiation dose received, usually 6 or 6.5 weeks);1, 3, 6, 12 months after the end of treatment
  Dysphagia is assessed by M.D.Anderson Dysphagia Inventory(score 20-100);Lower score indicates more severe symptoms
Quality of Life assessed by EORTC QLQ-C30 | 1 week before radiotherapy;at the middle of treatment(3 weeks after the start of radiotherapy);at the end of treatment(the last radiation dose received, usually 6 or 6.5 weeks);1, 3, 6, 12 months after the end of treatment
  Quality of Life is assessed by EORTC QLQ-C30(European Organization for Research and Treatment of Cancer Quality of Life Questionnaire);transformed into 0-100 scales for different domains and symptoms;Higher domain scores represent better quality of life, while higher symptom scores represent worse quality of life
Quality of Life assessed by QLQ-H&N35 | 1 week before radiotherapy;at the middle of treatment(3 weeks after the start of radiotherapy);at the end of treatment(the last radiation dose received, usually 6 or 6.5 weeks);1, 3, 6, 12 months after the end of treatment
  Quality of Life is assessed by QLQ-H&N35(Head and neck cancer-related quality of life scale);transformed into 0-100 scales for different domains and symptoms;Higher scores represent worse quality of life
Adverse effects | up to 12 months
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version(grade 1-5);Higher grade indicates more severe symptoms
Changes of oral flora | 1 week before radiotherapy;at the middle of treatment(3 weeks after the start of radiotherapy);at the end of treatment(the last radiation dose received, usually 6 or 6.5 weeks);1, 3, 6, 12 months after the end of treatment
  The changes of oral flora in patients' salivary or oral swab measured by 16s rDNA technique
Tongue range of motion | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Assessed by Tongue Range of Motion Assessment Scale(score 0-100);Lower score indicates more severe symptoms
Neck Fibrosis | 1 week before radiotherapy;weekly during the treatment(every 5 radiotherapy sessions);1, 3, 6, 12 months after the end of treatment
  Assessed by Common Terminology Criteria for Adverse Events (CTCAE) 5.0 version:Fibrosis skin(grade 1-5);Higher grade indicates more severe symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Xingchen Peng, Study Director — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China